CLINICAL TRIAL: NCT02308761
Title: A Dose Escalation Study of RO6870810/TEN-010 in Patients With Acute Myeloid Leukemia and Myelodysplastic Syndrome
Brief Title: A Study of RO6870810/TEN-010 in Participants With Acute Myeloid Leukemia and Myelodysplastic Syndrome
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NP39142
Record Dates: First submitted 2014-11-14; First posted 2014-12-04 (Estimated); Last update posted 2017-12-11 (Actual); Status verified 2017-12

CONDITIONS: Acute Myeloid Leukemia; Myelodysplastic Syndromes
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Myelodysplastic Syndromes | interventions — RO6870810

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- RO6870810 (Experimental): Participants with RR-AML and HMA-refractory MDS will receive RO6870810, as per schedule described in intervention description.
  Interventions: Drug: RO6870810

INTERVENTIONS:
Drug: RO6870810 — Participants will receive RO6870810 once daily (at escalated doses) via subcutaneous injection in either 28-day cycles (continuous 28 days dosing or 21 days dosing followed by 7 days off drug) or in 21-day cycle (14 days dosing followed by 7 days off drug), until MTD is identified.

SUMMARY:
RO6870810 (formerly TEN-010) is a small molecule, bromodomain and extra-terminal (BET) bromodomain inhibitor. This study is designed to characterize the safety, tolerability, and pharmacokinetics of RO6870810 monotherapy in participants with relapsed/refractory acute myeloid leukemia (RR-AML) and hypomethylating agent (HMA)-refractory myelodysplastic syndrome (MDS). The study will consist of a Screening Period, Treatment Period, and Post-Treatment Period. A standard 3+3 design will be used in which successive cohorts of three or more participants with RR-AML or HMA-refractory MDS will be treated at escalating doses until a maximum tolerated dose (MTD) is identiﬁed. Up to 51 adult participants with AML or MDS will be enrolled in the study.

ELIGIBILITY:
Inclusion Criteria:

* RR-AML
* Relapsed/refractory MDS
* Participants with a history of allogeneic stem cell transplant are eligible for study participation provided the following eligibility criteria are met:

  1. Transplant was more than (>) 100 days prior to study enrollment
  2. Participant has not taken immunosuppressive medications for at least 2 weeks
  3. No signs or symptoms of graft versus host disease other than Grade 1 skin involvement
  4. No active infection
* Eastern Cooperative Oncology Group Performance Status score equal to or less than (<=) 2
* Life expectancy of at least 2 months
* Disease-free of active second/secondary or prior malignancies for equal to or more than (>=) 1 year with the exception of currently treated basal cell or squamous cell carcinoma of the skin, or carcinoma in-situ of the cervix or breast
* Adequate hematological, renal, hepatic and coagulation laboratory test results
* Women of childbearing potential and men must agree to use adequate contraception from 28 days prior to the first dose of the study drug, during the entire Treatment Period, and for at least 28 days after the last dose of the study drug

Exclusion Criteria:

* New York Heart Association Class III or IV cardiac disease, myocardial infarction within the past 6 months, unstable arrhythmia
* Have Fridericia-corrected QT interval > 470 milliseconds (msec) (female) or > 450 msec (male), or history of congenital long QT syndrome
* Uncontrolled bacterial, viral, or fungal infections
* Known clinically important respiratory impairment
* Positive for human immunodeficiency virus, hepatitis B surface antigen, or hepatitis C antibodies
* History of major organ transplant
* Symptomatic central nervous system disease, malignancy, or metastasis
* Pregnant or nursing
* Concomitant chemotherapy, radiation therapy, immunotherapy, biologic therapy, or hormonal therapy
* Treatment with surgery or chemotherapy within 21 days prior to study entry
* Prior treatment with small molecule bromodomain and extra terminal family inhibitor
* Radiation for symptomatic lesions within 14 days of study enrollment
* Active substance abuse

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2014-11-06 (Actual); Primary Completion 2017-08-09 (Actual); Study Completion 2017-08-09 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants With Dose-Limiting Toxicities (DLTs) | Cycle 1 (cycle length = 21 or 28 days)
MTD of RO6870810 | Cycle 1 (cycle length = 21 or 28 days)
Percentage of Participants With Adverse Events (AEs) | Baseline up to 30 days after last dose (up to approximately 2.75 years)

SECONDARY OUTCOMES:
Area Under the Concentration Versus Time Curve from Time Zero to the End of Dosing Interval 24 Hours Later (AUC0-24) of RO6870810 | Cycle 1 Day 1 up to 2.75 years (detailed timeframe is provided in outcome description)
  Predose (Hour 0), immediately postdose and 0.25, 0.5, 1, 2, 4 hours postdose on Cycle 1 Day 1 and Cycle 1 Day 22 (Cycle 1 Day 22 is applicable only for 28-day continuous treatment); Predose (Hour 0), 4 hours postdose on Cycle 1 Day 2; Days 8, 15 of Cycle 1; Predose (Hour 0) on Day 1 of each treatment cycle from Cycle 2 up to end of treatment (approximately 2.75 years) (Cycle length = 21 or 28 days)
Maximum Observed Plasma Concentration (Cmax) of RO6870810 | Cycle 1 Day 1 up to 2.75 years (detailed timeframe is provided in outcome description)
  Predose (Hour 0), immediately postdose and 0.25, 0.5, 1, 2, 4 hours postdose on Cycle 1 Day 1 and Cycle 1 Day 22 (Cycle 1 Day 22 is applicable only for 28-day continuous treatment); Predose (Hour 0), 4 hours postdose on Cycle 1 Day 2; Days 8, 15 of Cycle 1; Predose (Hour 0) on Day 1 of each treatment cycle from Cycle 2 up to end of treatment (approximately 2.75 years) (Cycle length = 21 or 28 days)
Time to Cmax (Tmax) of RO6870810 | Cycle 1 Day 1 up to 2.75 years (detailed timeframe is provided in outcome description)
  Predose (Hour 0), immediately postdose and 0.25, 0.5, 1, 2, 4 hours postdose on Cycle 1 Day 1 and Cycle 1 Day 22 (Cycle 1 Day 22 is applicable only for 28-day continuous treatment); Predose (Hour 0), 4 hours postdose on Cycle 1 Day 2; Days 8, 15 of Cycle 1; Predose (Hour 0) on Day 1 of each treatment cycle from Cycle 2 up to end of treatment (approximately 2.75 years) (Cycle length = 21 or 28 days)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (2):
- United States (2):
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Weill Cornell Medical College, New York, New York

REFERENCES:
- [Derived] Roboz GJ, Desai P, Lee S, Ritchie EK, Winer ES, DeMario M, Brennan B, Nuesch E, Chesne E, Brennan L, Lechner K, Kornacker M, DeAngelo DJ. A dose escalation study of RO6870810/TEN-10 in patients with acute myeloid leukemia and myelodysplastic syndrome. Leuk Lymphoma. 2021 Jul;62(7):1740-1748. doi: 10.1080/10428194.2021.1881509. Epub 2021 Feb 13. PMID 33586590